CLINICAL TRIAL: NCT07007546
Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profile of Single or Multiple Oral Doses of ABSK061 Mini-tablets and to Evaluate the Effect of Soft Food With ABSK061 Mini-tablets on Its Pharmacokinetic Profile in Healthy Adult Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ABSK061 Mini-tablets in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABSK061-102
Record Dates: First submitted 2025-05-14; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single oral dose of ABSK061 (Experimental): Pharmacokinetic profile (PK) and safety of a single oral dose
  Interventions: Drug: ABSK061
- Multiple oral doses of ABSK061 (Experimental): The safety, tolerability, and PK profile of multiple oral doses of ABSK061
  Interventions: Drug: ABSK061
- Food Effect on ABSK061 (Experimental): Food Effect Tablet Formulation
  Interventions: Drug: ABSK061

INTERVENTIONS:
Drug: ABSK061 — A total of 18 healthy participants were planned to be enrolled in Part I and randomized 1: 1: 1 to Sequences A, B, and C. Participants in three sequences received a single dose of ABSK061 at doses of 1 mg, 10 mg, and 35 mg.
  Arms: Single oral dose of ABSK061
Drug: ABSK061 — A total of 12 healthy participants were planned to be enrolled in Part II, with multiple dose escalation trials prespecified in Sequences D and E, with 6 healthy participants in each sequence. In this MAD study, participants in Sequence D received ABSK061 microchips 5 mg QD(once a day) for 4 consecutive days.
  Arms: Multiple oral doses of ABSK061
Drug: ABSK061 — Part III plans to include 12 healthy participants randomized 1: 1: 1 to Sequence F, Sequence G, or Sequence H to receive a single oral dose of ABSK061 in triplicate doses of Treatment 1, Treatment 2, Treatment 3. Treatment 1 is 5 mg ABSK061 taken with 180 mL of water, Treatment 2 is 5 mg ABSK061 taken with a spoon of yogurt (approximately 15 mL), and Treatment 3 is administered with 5 mg ABSK061 with a spoon of applesauce (approximately 15 mL).
  Arms: Food Effect on ABSK061

SUMMARY:
To main objective is to evaluate the safety, tolerability, and pharmacokinetic profile of single or multiple oral doses of ABSK061 mini-tablets and to evaluate the effect of soft food with ABSK061 mini-tablets on its pharmacokinetic profile in healthy adult participants

ELIGIBILITY:
Inclusion Criteria:

* Gender:male or female participants, both male and female
* Age: 18 to 45 years (including 18 and 45 years)
* Weight: male participants weigh ≥ 50.0 kg, female participants weigh ≥ 45.0 kg, and body mass index is in the range of 19.0-26.0 kg/m2 (including cut-off value), and body mass index (BMI) = weight (kg)/height 2 (m2)
* Able to understand and willing to comply with the study procedures, voluntarily participate in this clinical trial and sign the informed consent form before screening

Exclusion Criteria:

* Significant history of any hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, immunologic, musculoskeletal disease, or allergic disease (as determined by the Investigator)
* Any ocular condition likely to increase the risk of eye toxicity
* Gastrointestinal disorders that will affect oral administration or absorption of ABSK061
* Females of child-bearing potential and males who plan to father a child while enrolled in this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-17 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics single-dose Cmax | Up to 48 hours post-dose
  maximum plasma concentration (Cmax)
Pharmacokinetics multiple-dose Cmax | Up to 24 hours post-dose
  maximum steady-state plasma concentration (Cmax)
Pharmacokinetics multiple-dose Cmin | Up to 24 hours post-dose
  average steady-state trough plasma concentration (Cmin)
Pharmacokinetics single dose Tmax | Up to 48 hours post-dose
  time to reach maximum plasma concentration (Tmax)
Pharmacokinetics single and multiple dose AUC | Up to 48 hours post-dose
  area under the plasma concentration-time curve (AUC)
Pharmacokinetics multiple-dose RAUC | Up to 24 hours post-dose
  accumulation ratio for AUC
Pharmacokinetics multiple-dose RCmax | Up to 24 hours post-dose
  accumulation ratio for Cmax (RCmax)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Initiation of study treatment up to 18-days post treatment
  number of participants with adverse events (AEs), serious adverse events (SAEs), as a measure of safety and tolerability
Number of participants with abnormal laboratory tests results and abnormal physical exam findings | Initiation of study treatment up to 18-days post treatment
  Frequency in changes in laboratory parameters and physical signs of toxicity

SECONDARY OUTCOMES:
Pharmacokinetics single dose CL/F | Up to 48 hours post-dose
  apparent total clearance (CL/F)
Pharmacokinetics single dose Vz/F | Up to 48 hours post-dose
  apparent volume of distribution (Vz/F)
Pharmacokinetics single dose t1/2 | Up to 48 hours post-dose
  half-life of ABSK061

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangnan University Affiliated Hospital, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-04-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT07007546/Prot_000.pdf